CLINICAL TRIAL: NCT03739437
Title: Automated Mobile Contingency Management for Smoking Cessation: A Pilot RCT
Brief Title: Automated Mobile Contingency Management for Smoking Cessation: A Pilot RCT (SCC PREVAILgo)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The wired carbon monoxide device (used to verify daily smoking abstinence) was discontinued by the manufacturer and replaced with a Bluetooth device which initially provided inaccurate readings.
Sponsor: University of Oklahoma (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9717; P30CA225520 (NIH)
Record Dates: First submitted 2018-10-25; First posted 2018-11-13 (Actual); Results first posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Smoking Cessation
Keywords: automated; smoking cessation; socioeconomic disadvantage; contingency management; financial incentives; mobile health; biochemical verification
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile Contingency Management (Experimental)
  Interventions: Behavioral: Mobile Contingency Management; Behavioral: Standard Care
- Standard Care (Active Comparator)
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Mobile Contingency Management — Participants will be offered six tobacco cessation telephone counseling sessions, 12 weeks of nicotine replacement therapy, and a smartphone app that remotely verifies participant identity and smoking abstinence and automatically credits a gift card account for evidence of smoking abstinence.
  Arms: Mobile Contingency Management
Behavioral: Standard Care — Participants will be offered six tobacco cessation telephone counseling sessions, 12 weeks of nicotine replacement therapy, and incentives that are not contingent on smoking abstinence (incentives are yoked to participants in the contingency management group).

SUMMARY:
The purpose of the proposed project is to pilot test an automated mobile phone-based contingency management (CM) approach to tobacco (smoking) cessation. With the assistance of the Mobile Health (mHealth) shared resource at the University of Oklahoma Health Sciences Center (OUHSC) and Stephenson Cancer Center (SCC), the investigators have combined technologies including 1) low-cost carbon monoxide monitors that connect with mobile phones to remotely verify smoking abstinence, 2) facial recognition software to confirm the identity of participants while they provide a breath sample, and 3) remote delivery of incentives automatically triggered by biochemical confirmation of self-reported smoking abstinence. This automated, mobile CM approach will be evaluated in a randomized controlled pilot trial of 40 socioeconomically disadvantaged males and females seeking smoking cessation treatment. Participants will be randomly assigned to telephone counseling plus nicotine replacement therapy (standard care [SC]) or SC plus a 12-week mobile financial incentives intervention (CM) for biochemically-confirmed abstinence. Participants will be followed for 12 weeks after a scheduled quit attempt to assess smoking status.

DETAILED DESCRIPTION:
Tobacco Cessation Treatment. Participants referred to the Tobacco Treatment Research Program (TTRP) for smoking cessation treatment who are interested and eligible for the current study will be offered weekly telephone counseling/support sessions led by a staff counselor. Six unique sessions covering the following topics will be offered: 1) quit planning 2) the impact of tobacco on health/benefits of quitting, 2) stress management strategies, 3) making positive lifestyle changes, 4) developing coping skills, and 5) relapse prevention. The counselor will check in with participants each week about the difficulties and successes they have experienced, and plan for any challenging situations that are anticipated. Advice and support will be provided as needed. A two-week supply of nicotine replacement therapy (patches and gum) will be offered during the first session for medically eligible participants. Additional patches and gum will be mailed out for participants who wish to continue using pharmacotherapy (for up to 12 weeks).

Financial Incentives. Participants will be provided with a smartphone that has the SCC PREVAILgo EMA app preloaded, as well as a Smokerlyzer iCO monitor. Participants will be randomly prompted 4 times daily during waking hours to complete smartphone-based EMAs (ecological momentary assessments). During random prompts, participants who self-report abstinence will be asked to provide a CO breath sample on 5 randomly selected days out of the week. Participants will be prompted to provide a CO breath sample at the last random assessment of the day, Participants will be reminded 2 additional times on the same day during their normal waking hours to provide a CO breath sample if they miss the initial assessment. A gift card credit may be earned following a self-report of abstinence during the past 24 hours combined with a breath CO sample of ≤ 6 ppm.

Recruitment/Screening (Visit 1, Part 1; Screening). Individuals who are referred to the TTRP for smoking cessation treatment and report that they are uninsured or receiving Medicaid benefits will be sent an informational handout with their TTRP information packet (prior to their first visit). Participants will be reminded of all future in-person appointments via telephone, mail, email, and/or text. Additionally, research staff may attempt to collect smoking cessation status with each reminder. Participants with transportation difficulties living in the Oklahoma City metro area may be scheduled for pick-up and drop-off for key visits with SendaRide through their secure dashboard. At the first visit, study staff will inquire about their interest in finding out more about the study. Study staff will review the consent form with interested participants, and they will be screened for eligibility on-site in a private room in the clinic. Participant eligibility for the current study will not influence eligibility for the TTRP. The Rapid Estimate of Adult Literacy in Medicine (REALM; see Appendix A) will be administered to ensure that all participants are able to read at ≥ sixth grade level (i.e., required to complete EMA and self-report questionnaires). Expired carbon monoxide (CO) will be measured and participants will be questioned about their 1) insurance status 2) age, 3) current level of smoking, 4) willingness to quit smoking, 5) willingness/ability to complete 6 weekly counseling sessions (including the first visit), 6) pregnancy/breastfeeding status, 7) computer/internet access, and 8) contraindications for nicotine replacement therapy. Expired CO will be measured. Eligible participants may complete the assessment portion of the visit.

Pre-Quit (Visit 1, Part 2; Assessment). Participants will complete self-report questionnaires on a laptop computer; weight and height will be measured in a private room to ensure confidentiality. Visit 1 will be 1 of 2 in-person visits. Participants will be provided with an Android smartphone and a Smokerlyzer iCO breathe monitor. They will be instructed regarding the use of the phone (participants may make personal calls), the EMA procedures, and use of the portable CO monitor. Participants will receive 4 random prompts and 1 daily diary prompt (in the morning) during the normal waking hours each day for five consecutive weeks. Participants will be instructed to quit smoking at bedtime or 10:00 pm (whichever occurs first) 7 days after enrollment.

Quit Day. Participants will remotely complete web-based self-report questionnaires and provide a smartphone-based CO measurement.

One Week Post-Quit. Participants will remotely complete web-based self-report questionnaires and provide a smartphone-based CO measurement.

Two Weeks Post-Quit. Participants will remotely complete web-based self-report questionnaires and provide a smartphone-based CO measurement.

Three Weeks Post-Quit. Participants will remotely complete web-based self-report questionnaires and provide a smartphone-based CO measurement.

Four Weeks Post-Quit. Participants will remotely complete web-based self-report questionnaires and provide a smartphone-based CO measurement.

Eight Weeks Post-Quit. Participants will remotely complete web-based self-report questionnaires and provide a smartphone-based CO measurement.

Twelve Weeks Post-Quit. Participants will return to the TTRP and complete self-report questionnaires on a tablet or laptop computer and provide a CO measurement.

ELIGIBILITY:
1. annual Household income of < 200% of the federal poverty threshold (i.e., low-income) given household size
2. earn a score ≥ 4 on the REALM indicating > 6th grade English literacy level
3. are willing to quit smoking 7 days after enrollment
4. are ≥ 18 years of age
5. currently smoke ≥ 5 cigarettes per day
6. have a CO level of > 6 ppm
7. have no contraindications for NRT
8. willingness to complete an identity check (i.e., video conference call or provide a photo ID).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darla Kendzor, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile Contingency Management | Standard Care
Started | 9 | 11
Completed | 7 | 6
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Contingency Management | Standard Care | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.33 (10.04) | 57.45 (8.39) | 55.60 (9.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 11 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported Smoking Cessation
Description: Self-reported smoking abstinence during the past 7 days days
Time Frame: 13 weeks post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Contingency Management | Standard Care
Number analyzed (Participants) | 9 | 11
Participants | 4 | 2
Statistical Analysis 1: Comparison: Mobile Contingency Management vs Standard Care; Test type: Superiority; p = 0.384, Chi-squared

2. Primary Outcome: Completion of Breath Sample Submissions
Description: The percentage of total possible smartphone-based breath sample submissions completed over 13 weeks.
Time Frame: 13 weeks post-enrollment
Measure: Number; unit: Breath samples submitted
Units Other Than Participants: Total Possible Breath Sample Submissions
Arm/Group | Mobile Contingency Management | Standard Care
Number analyzed (Participants) | 9 | 11
Number analyzed (Total Possible Breath Sample Submissions) | 819 | 1001
Breath samples submitted | 422 | 566

3. Secondary Outcome: Loss of Smartphones
Description: The total number of smartphones lost by participants during the study.
Time Frame: 13 weeks post-enrollment
Population: A total of 9 phones were provided to participants (all other participants used their own phones).
Measure: Number; unit: Number of phones lost
Arm/Group | Mobile Contingency Management | Standard Care
Number analyzed (Participants) | 5 | 4
Number of phones lost | 2 | 1

4. Secondary Outcome: Loss of iCO Sensors
Description: The total number of iCO Sensors lost by participants during the study.
Time Frame: 13 weeks post-enrollment
Measure: Number; unit: Number of iCOs lost
Arm/Group | Mobile Contingency Management | Standard Care
Number analyzed (Participants) | 9 | 11
Number of iCOs lost | 2 | 0

ADVERSE EVENTS:
Time Frame: Participants were followed for 13 weeks post-enrollment (1 week pre-quit-date through 12 weeks post-quit-date).
Arm/Group | Mobile Contingency Management | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT03739437/Prot_000.pdf
  • Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT03739437/ICF_001.pdf